CLINICAL TRIAL: NCT00331097
Title: Adjuvant Chemotherapy in Elderly Patients With Breast Cancer: Weekly Docetaxel vs. CMF
Brief Title: ELDA: Elderly Breast Cancer - Docetaxel in Adjuvant Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELDA
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: elderly; adjuvant therapy; intermediate risk; high risk
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Methotrexate; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Standard chemotherapy with CMF
  Interventions: Drug: cyclophosphamide; Drug: methotrexate; Drug: 5-fluorouracil
- B (Experimental): Weekly docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — 35 mg/m2 intravenously on days 1, 8, and 15 every 28 days
  Arms: B
Drug: cyclophosphamide — 600 mg/m2 intravenously days 1, 8 every 28 days
  Arms: A
Drug: methotrexate — 40 mg/m2 intravenously days 1 and 8 every 28 days
  Arms: A
Drug: 5-fluorouracil — 600 mg/m2 intravenously days 1 and 8 every 28 days
  Arms: A

SUMMARY:
The purpose of this study is to compare disease free survival of elderly breast cancer patients treated with standard adjuvant chemotherapy (CMF) versus experimental adjuvant chemotherapy (weekly docetaxel).

DETAILED DESCRIPTION:
Adjuvant combination chemotherapy, given after breast cancer surgery, has been established as the standard approach to reduce the risk of breast cancer recurrence in those patients at intermediate or high risk for recurrence. However, since elderly patients have been underrepresented in past clinical trials, the optimal adjuvant therapy for elderly patients at risk for recurrence has not yet been defined.

Docetaxel is one of the most active drugs for patients with metastatic breast cancer and several trials are evaluating its efficacy in the adjuvant setting. Administration of docetaxel on a weekly schedule is effective and well tolerated in women with metastatic breast cancer.

In this study, patients from ages 65 to 80 will be randomized to one of two treatment strategies:

* standard adjuvant chemotherapy with CMF (cyclophosphamide, methotrexate, and 5-fluorouracil given intravenously on days 1 and 8 of each cycle)
* experimental adjuvant chemotherapy with weekly docetaxel (given intravenously on days 1,8, and 15 of each cycle)

In both treatment strategies:

* 4 cycles of chemotherapy will administered for patients at least 10% positive for ER or PgR, and 6 cycles will administered for patients expressing < 10% ER or PgR
* patients with any positive expression of ER or PgR will receive adjuvant hormonal therapy with tamoxifen (20mg/day for 5 years) after concluding chemotherapy
* adjuvant radiation therapy will be given to patients who are candidates at the conclusion of chemotherapy and within 6 months of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive unilateral breast cancer
* Age > 65 and < 80 years
* Intermediate-high risk of recurrence according to St. Gallen criteria: ER negative and PgR negative, or axillary lymph node metastasis, or tumor size > 2 cm, or tumor grade 2 or 3 (intermediate or high)

Exclusion Criteria:

* Performance status >1
* Distant metastasis
* Concomitant malignancy or malignancy within previous 5 years (except basal cell or spinocellular skin cancer and in situ cervical cancer if they have been adequately treated
* Previous breast cancer treatment
* Neutrophils < 2000/mm3 or platelets < 100000/mm3 or haemoglobin < 10 g/dl
* Creatinine > 1.25 the upper normal limit
* GOT and-or GPT and/or bilirubin > 1.25 the upper normal limit
* Concomitant conditions that contraindicate the use of the drugs in the protocol
* Incapacity or refusal to provide informed consent

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2003-07; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
disease free survival | at 5 years

SECONDARY OUTCOMES:
toxicity | weekly
compliance | every 3 weeks
quality of life | baseline and every 3 weeks during therapy
overall survival | at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Giuseppe D'Aiuto, M.D., Principal Investigator — NCI Naples, Division of Surgical Oncology A; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (8):
- Italy (8):
  - Azienda Sanitaria S. Giuseppe Moscati, Monteforte Irpino, AV
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Policlinico Monteluce, Sant'Andrea Delle Frate, PG
  - Azienda Ospedaliera Cardarelli, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli
  - Università Federico II, Cattedra di Oncologia Medica, Napoli
  - Az. Osp. Treviglio - Caravaggio, Treviglio
  - Ospedale S. Luca ASL SA 3, Vallo della Lucania

REFERENCES:
- [Background] Nuzzo F, Morabito A, De Maio E, Di Rella F, Gravina A, Labonia V, Landi G, Pacilio C, Piccirillo MC, Rossi E, D'Aiuto G, Thomas R, Gori S, Colozza M, De Placido S, Lauria R, Signoriello G, Gallo C, Perrone F, de Matteis A. Weekly docetaxel versus CMF as adjuvant chemotherapy for elderly breast cancer patients: safety data from the multicentre phase 3 randomised ELDA trial. Crit Rev Oncol Hematol. 2008 May;66(2):171-80. doi: 10.1016/j.critrevonc.2007.10.006. Epub 2007 Dec 21. PMID 18160303
- [Result] Perrone F, Nuzzo F, Di Rella F, Gravina A, Iodice G, Labonia V, Landi G, Pacilio C, Rossi E, De Laurentiis M, D'Aiuto M, Botti G, Forestieri V, Lauria R, De Placido S, Tinessa V, Daniele B, Gori S, Colantuoni G, Barni S, Riccardi F, De Maio E, Montanino A, Morabito A, Daniele G, Di Maio M, Piccirillo MC, Signoriello S, Gallo C, de Matteis A. Weekly docetaxel versus CMF as adjuvant chemotherapy for older women with early breast cancer: final results of the randomized phase III ELDA trial. Ann Oncol. 2015 Apr;26(4):675-682. doi: 10.1093/annonc/mdu564. Epub 2014 Dec 8. PMID 25488686
- [Derived] Di Maio M, Gallo C, Leighl NB, Piccirillo MC, Daniele G, Nuzzo F, Gridelli C, Gebbia V, Ciardiello F, De Placido S, Ceribelli A, Favaretto AG, de Matteis A, Feld R, Butts C, Bryce J, Signoriello S, Morabito A, Rocco G, Perrone F. Symptomatic toxicities experienced during anticancer treatment: agreement between patient and physician reporting in three randomized trials. J Clin Oncol. 2015 Mar 10;33(8):910-5. doi: 10.1200/JCO.2014.57.9334. Epub 2015 Jan 26. PMID 25624439